CLINICAL TRIAL: NCT02452853
Title: Hepatic Resection Combined With or Without Oxaliplatin+5-Fluorouracil/ Leucovorin(5-FU/LV)(FOLFOX4) for Resectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Brief Title: HR Combined With FOLFOX4 for HCC With PVTT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, M.D.,Ph.D., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC002
Record Dates: First submitted 2015-05-05; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HR combined with FOLFOX4 (Experimental): 1. HR ;
  2. FOLFOX4 4 weeks after HR
  Interventions: Procedure: HR; Drug: FOLFOX4

INTERVENTIONS:
Procedure: HR — HR:
  HR was carried out under general anesthesia using a right subcostal incision with a midline extension. Intraoperative ultrasound was routinely performed. Pringle's maneuver was routinely used with a clamp/unclamp time of 10 minutes/5 minutes.Thrombectomy was performed according to the location and extent of PVTT. The en bloc technique was used for patients if the portal vein branch could be ligated with a sufficient safety margin between its root and the tip of the thrombus
Drug: FOLFOX4 — FOLFOX4(Oxaliplatin + 5-Fluorouracil/Leucovorin):
  4 weeks after HR; Drug: Oxaliplatin + 5- Fluorouracil/Leucovorin Day 1: Oxaliplatin 85mg/m² 2h IV infusion, leucovorin 200mg/m² 2h IV infusion, 5-fluorouracil 400mg/m² IV bolus, 5-fluorouracil 600mg/m2 22h IV infusion.
  Day 2: Leucovorin 200mg/m² 2h IV infusion, 5-fluorouracil 400mg/m² IV bolus, 5-fluorouracil 600mg/m² 22h IV infusion. Repeated every 2 weeks

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most common cancer and the third most frequent cause of cancer death worldwide. Hepatic resection (HR) is the conventional ''curative'' treatment for HCC. In both the European and the United States Proposed Guidelines for HCC, HR is recommended only for patients with preserved liver function and with early stage HCC. Unfortunately, because of tumor multifocality, portal vein invasion, and underlying advanced cirrhosis, only 10% to 30% of HCCs are amenable to such a ''curative'' treatment at the time of diagnosis. Transarterialchemoembolization (TACE) has become the most popular palliative treatment for patients with unresectable HCC, and it is no longer considered as a contraindication to HCC with portal vein tumor thrombus (PVTT). Unfortunately, the long-term outcomes are generally poor for HCC treated with TACE, especially for HCC with PVTT. To improve on the results of treatment of HCC with PVTT, attempts have been made to perform HR for these patients. HCC with PVTT remains a contraindication to liver transplantation because of the high rate of tumor recurrence, and because of the severe shortage of donor organs. HR remains the only therapeutic option that may still offer a chance of cure. With advances in surgical techniques, it has become feasible to remove all gross tumors, including PVTT, which has extended to the main portal vein, safely by surgery. More HCC with PVTT, which previously were considered as unresectable, have become resectable.Recent studies have even shown favorable long-term survival outcomes of HR in well-selected cases of HCC with PVTT. However, the recurrence rate after HR for PVTT is still high and the prognosis for patients with HCC with PVTT is very poor. Systemic chemotherapy is considered to be one of the main treatments for malignant tumors. HCC is known to be highly refractory to conventional systemic chemotherapy because of its heterogeneity and multiple etiologies. Before the advent of the molecular-targeted agent sorafenib, which has subsequently become the standard of care, no standard systemic drug or treatment regimen had shown an obvious survival benefit in HCC. Nowadays, there is no systemic chemotherapy regimen had been definitively recommended as the standard for treating HCC. Clinical activity of several regimens containing oxaliplatin (OXA) in advanced HCC had been demonstrated in phase II studies. In a phase II study of the FOLFOX4 (infusional fluorouracil [FU], leucovorin[LV], and OXA) regimen in Chinese patients with HCC, median overall survival (OS) was 12.4 months, mean time to progression was 2.0 months, and the response rate (RR) was 18.2%. The safety profile was acceptable. Recently, the results of a phase Ⅲ randomize study showed that FOLFOX4 served as palliative chemotherapy can induce higher overall survival, progression-free survival and response rate comparing to doxorubicin in patients with advanced hepatocellular carcinoma from Asia. The safety data was also acceptable.So the investigators' hypothesis is that post-surgery FOLFOX4 can reduce high recurrence rate after HR for HCC with PVTT. The aim of this open-label, single prospective study is to evaluate the efficacy and safety of HR combined with FOLFOX4 systemic chemotherapy for patients with HCC with PVTT.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years;
2. Presence of PVTT on imaging, except PVTT extending to involve the superior mesenteric vein
3. ECOG status 0;
4. Resectable disease( defined as the possibility of completely removing all gross tumors and retaining a sufficient liver remnant to sustain life)

Exclusion Criteria:

1. the presence of extrahepatic spread on imaging;
2. a Child-Pugh class C liver cirrhosis, or ICG-R15 >30%, or evidence of hepatic decompensation including ascites, esophageal, or gastric variceal bleeding or hepatic encephalopathy;
3. an American Society of Anesthesiologists (ASA) score ≥3.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2 years
Number of Complications reported using the National Cancer Institute Common Toxicity Criteria grading version 4.0 | 2 years

SECONDARY OUTCOMES:
Recurrence-free survival | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, M.D.,Ph.D., Study Chair — Sun Yat-sen University

REFERENCES:
- [Background] Peng ZW, Guo RP, Zhang YJ, Lin XJ, Chen MS, Lau WY. Hepatic resection versus transcatheter arterial chemoembolization for the treatment of hepatocellular carcinoma with portal vein tumor thrombus. Cancer. 2012 Oct 1;118(19):4725-36. doi: 10.1002/cncr.26561. Epub 2012 Feb 22. PMID 22359112
- [Background] Qin S, Bai Y, Lim HY, Thongprasert S, Chao Y, Fan J, Yang TS, Bhudhisawasdi V, Kang WK, Zhou Y, Lee JH, Sun Y. Randomized, multicenter, open-label study of oxaliplatin plus fluorouracil/leucovorin versus doxorubicin as palliative chemotherapy in patients with advanced hepatocellular carcinoma from Asia. J Clin Oncol. 2013 Oct 1;31(28):3501-8. doi: 10.1200/JCO.2012.44.5643. Epub 2013 Aug 26. PMID 23980077